CLINICAL TRIAL: NCT03537001
Title: Use of Inhaled Methoxyflurane (Penthrox®) as an Analgesic in Extra-hospital Traumatology at EMS37
Brief Title: Use of Penthrox in Extra-hospital Traumatology
Acronym: UPETEH
Status: Completed | Type: Observational
Sponsor: University Hospital, Tours (Other)
Responsible Party: Sponsor
Other Study IDs: RIPH3-RNI17/UPETEH; 2017-A01077-46 (Other: IdRCB)
Record Dates: First submitted 2018-04-25; First posted 2018-05-25 (Actual); Last update posted 2019-04-24 (Actual); Status verified 2019-04

CONDITIONS: Pain, Acute; Trauma Injury; Pain Management
Keywords: Methoxyflurane; Penthrox; anesthetic; analgesia; acute; traumatic; pain; prehospital setting; visual numeric scale
MeSH Terms: conditions — Acute Pain; Accidental Injuries; Agnosia; Pain

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Penthrox: Administration of Penthrox at the beginning of the management of the traumatized adult patient
  Interventions: Other: Penthrox

INTERVENTIONS:
Other: Penthrox — Self-administration of penthrox by the patient under the supervision of a physician trained in its administration, in strict compliance with its MA.

SUMMARY:
In pre-hospital settings, the administration of analgesics is often delayed because of difficult patient access (incarceration), difficulty finding a venous pathway or patient refusal.

An optimization of the management of pain in urgency is therefore still necessary.

A side from nitrousoxide of which usage remains restrictive, methoxyflurane (Penthrox®) is the only volatile analgesic currently available for pre-hospital use.

The purpose of this study is to answer the question: Does the use of the inhaled route with Penthrox add value to the treatment of acute traumatic pain in the pre-hospital stage?

DETAILED DESCRIPTION:
In pre-hospital settings, the administration of analgesics is often delayed because of difficult patient access (incarceration), difficulty finding a venous pathway or patient refusal.

An optimization of the management of pain in urgency is therefore still necessary.

A side from nitrousoxide of which usage remains restrictive, methoxyflurane (Penthrox®) is the only volatile analgesic currently available for pre-hospital use.

Methoxyflurane (Penthrox®) is a single-use inhalation non-opioid analgesic for the management of moderate to severe traumatic pain. This treatment has been used in New Zealand and Canada for over 20 years for the management of acute pain in adults and children. It was granted marketing authorization in Europe in 2016 and has been marketed in France since 2017.

The purpose of this study is:

* To study the efficacy and safety of Penthrox, administrated at the beginning of the management of the traumatized adult patient.
* Assess the comfort of patients and caregivers
* To answer the question: Does the use of the inhaled route with Penthrox add value to the treatment of acute traumatic pain in the pre-hospital stage?

ELIGIBILITY:
Inclusion Criteria:

* Conscious Patient
* Age ≥ 18 years
* Acute pain only of traumatic origin
* Pain > 4 on a visual numerical scale (VNS)
* Stable hemodynamic conditions (PA> 90/60)

Non Inclusion Criteria:

* Pregnant or nursing woman
* Patient who has already received analgesics
* Patient benefiting from an intravenous approach for analgesia
* Known renal or hepatic disease
* Hypersensitivity to fluorinated anesthetics or history of malignant hyperthermia of the patient or family.
* Respiratory distress
* Patient who objected to the processing of his data

Exclusion Criteria:

* Intravenous injection for analgesia

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients treated by the ER at Tours hospital which correspond to the inclusion, non-inclusion & exclusion criterias.
Sampling Method: Non-Probability Sample
Enrollment: 20 (Actual)
Dates: Start 2017-08-29 (Actual); Primary Completion 2018-08-30 (Actual); Study Completion 2018-08-30 (Actual)

PRIMARY OUTCOMES:
Change of traumatic acute pain level between baseline and 5 minutes | Baseline, 5 minutes
  Efficiency will be measured by its effect on pain according to a visual numerical scale (VNS: between 0 and 10).

SECONDARY OUTCOMES:
Change of traumatic acute pain level between baseline and 10 minutes | Baseline, 10 minutes
  Efficiency will be measured by its effect on pain according to a visual numerical scale (VNS: between 0 and 10).
Pain extinction duration | Baseline, 10 & 15 minutes
  Duration before pain extinction, evaluated using a visual numerical scale (VNS: between 0 and 10) at 0, 10 & 15 minutes.
Penthrox tolerance | Through study completion, an average of 30 minutes
  Collection of side effects
Medical team level of satisfaction | 30 minutes
  5 grades satisfaction scale filled by the medical team 30 minutes after the treatment (Very satisfied, Satisfied, Neutral, Dissatisfied, Very dissatisfied)
Patient level of satisfaction | 30 minutes
  5 grades satisfaction scale filled by the patient 30 minutes after the treatment (Very satisfied, Satisfied, Neutral, Dissatisfied, Very dissatisfied)
Change of traumatic acute pain level between 0 and15 minutes | Baseline, 15 minutes
  Efficiency will be measured by its effect on pain according to a visual numerical scale (VNS: between 0 and 10).

CONTACTS AND LOCATIONS:
Overall Officials: Sanaa El Azhari, MD, Principal Investigator — sanaa.elazari@gmail.com
Locations (1):
- Emergency Medical Service, University Hospital, Tours, Tours, France

IPD SHARING:
Plan to Share IPD: No